CLINICAL TRIAL: NCT06905561
Title: Topical Diclofenac for Prevention of Radiation-induced Dermatitis: A Single-center, Randomized Controlled Trial
Brief Title: Topical Diclofenac for Prevention of Radiation-induced Dermatitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Hainan Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2025-K01-01
Record Dates: First submitted 2025-02-07; First posted 2025-04-01 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-02

CONDITIONS: Head and Neck Tumor; Breast Cancer
Keywords: Topical Diclofenac; Radiation-induced dermatitis; Prevention; Head and Neck tumor; Brest Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Breast Neoplasms; Radiodermatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group（diclofenac sodium gel ） (Experimental): In addition to routine skin care, diclofenac sodium gel was applied to the skin of the irradiated site triple a day a day from the date of first radiotherapy until end of radiotherapy or until the test side skin developed ≥grade 3 RID.Conventional health care:Minimize skin irritation, friction and excessive sun exposure in the irradiated area (level III to IV evidence), avoid wearing high-neck and tight clothing, and recommend low-neck tops. Subjects wash irradiated skin with water or wet towel, and wipe skin with dry towel to keep irradiated skin clean and dry.
  Interventions: Drug: Diclofenac Sodium Gel
- control group（Placebo Comparator） (Placebo Comparator): In addition to routine skin care, Placebo gel was applied to the skin of the irradiated site triple a day a day from the date of first radiotherapy until end of radiotherapy or until the test side skin developed ≥grade 3 RID.Conventional health care:Minimize skin irritation, friction and excessive sun exposure in the irradiated area (level III to IV evidence), avoid wearing high-neck and tight clothing, and recommend low-neck tops. Subjects wash irradiated skin with water or wet towel, and wipe skin with dry towel to keep irradiated skin clean and dry.
  Interventions: Other: Placebo gel

INTERVENTIONS:
Drug: Diclofenac Sodium Gel — Diclofenac Sodium Gel were applied to the skin of the irradiated site triple a day a day from the date of first radiotherapy until end of radiotherapy or until the test side skin developed ≥grade 3 RID.
  Arms: Treatment group（diclofenac sodium gel ）
Other: Placebo gel — The placebo does not contain the active ingredients of Jalosome, only the co-formulants.
  Arms: control group（Placebo Comparator）

SUMMARY:
Radiation induced dermatitis (RID) is one of the leading adverse events of radiation therapy, and if occurred could alter the course of therapy. The main pathways of RID is inflammation and oxidative stress on local and systemic bases. The Diclofenac is a COX-2 inhibitor and Nonsteroidal anti-inflammatory drugs whose anti-inflammatory and antioxidant activities have been proven in several clinical trials. Thus, the aim of the present study is to evaluate the efficacy of Diclofenac sodium gel as a prophylactic method against the development of RID.

DETAILED DESCRIPTION:
Radiation induced dermatitis (RID) is one of the most commonly reported adverse events of Head and neck tumor, breast cancer radiation therapy (RT). Radiation therapy toxicity is exhibited within hours to weeks of exposure and persisting throughout the course of treatment. Radiation induced dermatitis is a result of generation of reactive oxygen species (ROSs), which in return induces epidermal and dermal inflammatory responses. Radiation causes structural tissue damage, which trigger production of pro-inflammatory mediators; as NF-κB, COX-2, and cytokines such as IL-6, TNF-a, and IFN- γ. Subsequently erythema, ulceration, and edema are developed，then followed by thinning of the epidermis, dry desquamation. If damage is more severe, moist desquamation occur. It can be deduced that inflammatory response plays a significant role in the radiotherapy induced dermatitis.

There are many agents that are used in the management of RID in the clinical settings, however, up till now there is none supported by the guidelines. Radiation induced dermatitis occurrence, not only could it impair the patient's quality of life but it could also affect the RT course of treatment, which could negatively influence the cancer treatment. Therefore more effort is needed to find a method of prevention of RID, resulting from Head and neck tumor,breast cancer RT.

Diclofenac sodium gel, a COX-2 inhibitor and nonsteroidal anti-inflammatory drug (non-NSAID), is widely used to treat inflammatory conditions, and studies show that topical diclofenac has no safety concerns. It has been used for more than 20 years in patients with osteoarthritis without any significant adverse effects. The combination of diclofenac sodium as a COX-2 inhibitor and ionising radiation not only enhances the effect of radiation on tumour cells, but also improves radiation therapy for patients. Studies have shown that diclofenac sodium gel, through COX-2, can be used to prevent the development of capecitabine-induced hand-foot syndrome (HFS). RID upregulates COX-2 due to inflammatory stimulation, and COX-2 indirectly produces reactive oxygen species (ROS). The investigators conclude that diclofenac gel can reduce ROS by locally inhibiting COX-2 enzyme, thus preventing radiation dermatitis and reducing skin damage. Therefore, the investigators plan to conduct a study on the use of diclofenac sodium gel in radiation dermatitis to investigate the incidence of RID grade 2 and above at different time points after radiotherapy in patients with head and neck tumours, and whether it can reduce the incidence and severity of RID-related symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female which are 18 years of age or older
2. Performance status < 2
3. Epithelial carcinoma of oropharynx, nasopharynx, larynx, hypopharynx, paranasal sinus and salivary glands or breast cancer, planned to receive a total dose of at least 50 Gy
4. The RTOG radiation dermatitis rating should be equal to 0 and the skin nutrition should be good
5. The main organs are functioning normally and meet the following standards: (1) Blood routine examination must meet the following criteria: (no blood transfusion within 14 days) a. HB ≥ 100g/L, b. WBC ≥3×10^9/L c. ANC≥1.5×10^9/L, d. PLT ≥100×10^9/L; (2) Biochemical examination must meet the following standards: a. BIL<1.5 times the upper limit of normal value (ULN), b. ALT and AST<2.5ULN, GPT ≤1.5×ULN; c. Serum Cr≤1 ULN, endogenous creatinine clearance rate>60ml/min (Cockcroft Gault formula);(3).Good coagulation function: defined as International standardized ratio (INR) or prothrombin time (PT) ≤1.5×ULN;(4).The myocardial enzyme spectra were in the normal range.
6. Patients willing and able to give signed informed consent and, in the opinion of the Investigator, to comply with the Clinical Investigation Plan tests and procedures.

Exclusion Criteria:

1. Pregnant or lactating women
2. A known history of intolerance or allergy to any component of the investigational product;
3. severe cardiopulmonary disease (such as unstable angina attacks, grade II cardiac insufficiency, acute myocardial infarction, acute episodes of chronic obstructive pulmonary disease, pulmonary heart disease);
4. The acute phase is accompanied by inflammatory skin diseases, such as atopic dermatitis, contact dermatitis, psoriasis, lichen planus, pityriasis rosea.
5. Systemic diseases known to delay the skin healing process, such as diabetes or severe kidney failure;
6. Skin rupture caused by malignant tumors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of development of grade ≥ 2 RID | From the first day of radiotherapy until 2 weeks after the end of radiotherapy
  If the patient developed grade ≥ 2 RID or not, RTOG standards were used for evaluation

SECONDARY OUTCOMES:
Evaluation of Time to develop grade ≥2 RID | From the first day of radiotherapy until 2 weeks after the end of radiotherapy
  EvaluationTime to develop grade ≥ 2 RID incidence, will be assessed by RTOG criteria based on the clinical presentation of Time to develop grade ≥2 RID
Evaluation of Pain Intensity | From the first day of radiotherapy until 2 weeks after the end of radiotherapy
  Pain related assessment will be done through a Visual Analog Scale, with 0 being No pain and 10 being unbearable pain
Evaluation of Incidence of Treatment-Emergent Adverse Events | From the first day of radiotherapy through treatment completion(up to 7 weeks or 5 weeks)
  Patients will be educated and instructed to report any adverse events
Evaluation of Quality of life | From the first day of radiotherapy until 2 weeks after the end of radiotherapy
  Skin-related quality of life assessed through the Dermatology Life Quality Index (DLQI)
Incidence of radiotherapy interruption | From the first day of radiotherapy through treatment completion (up to 7 weeks or 5 weeks)
  If the patient has been interrupted by RID or not
The Concentration of inflammatory factors (IL-2、IL-4 、IL-6、IL-10、interferon-γ、TNF-α) | Baseline（Day 0） and through study completion（Day 36 or Day 46）
  The differences in expression of inflammatory factors, such as IL-2 (pg/ml）,IL-4 (pg/ml）,IL-6 (pg/ml）,IL-10 (pg/ml）,interferon-γ（pg/ml） and TNF-α（pg/ml）.
The Concentration of inflammatory factors (WBC) | Baseline（Day 0） and through study completion（Day 36 or Day 46）
  The differences in expression of inflammatory factors, such as WBC(10^9/L).
The Concentration of inflammatory factors (CRP) | Baseline（Day 0） and through study completion（Day 36 or Day 46）
  The differences in expression of inflammatory factors, such as CRP（mg/L）.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Hainan Medical University, Haikou, Hainan, China